CLINICAL TRIAL: NCT01034839
Title: Role of Consolidation With High-dose Cytarabine in Overall Survival of Adults With Acute Myeloid Leukemia
Brief Title: High-dose Cytarabine and Survival in AML
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Murilo Chermont Azevedo, University of Sao Paulo, General Hospital
Other Study IDs: mcazevedo01
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; prognosis; cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute myeloid leukemia, adults: Adults treated for acute myeloid leukemia in our hospital between 1978 and 2007

SUMMARY:
In adults with acute myeloid leukemia, especially those < 60 years of age, high-dose cytarabine consolidation therapy has been shown to influence survival, but the appropriate dose has not been defined.

DETAILED DESCRIPTION:
Background In adults with acute myeloid leukemia, especially those < 60 years of age, high-dose cytarabine consolidation therapy has been shown to influence survival. However, the appropriate dose has not been defined. We evaluated survival after cytarabine consolidation therapy at three different doses.

Design and Methods We conducted a single-center, retrospective study involving 499 acute myeloid leukemia patients, aged 18-92 years, all evaluated between 1978 and 2007. Of those 499 patients, 400 received curative treatment and 203 received cytarabine consolidation. The latter were divided into three groups: low-dose (receiving < 1.5 g/m2 of i.v. cytarabine, every 12 h, on 3 alternate days, for up to 4 cycles); medium-high-dose (< 45.45 g-the median dose-by the end of the cycles); and very-high-dose (≥ 45.45 g by the end of the cycles).

Results Among the 400 patients receiving curative treatment, five-year survival was 22.8% (91 patients). Cytarabine consolidation dose was an independent determinant of survival (significant differences were found among the groups), whereas age, karyotype, induction protocol, French-American-British classification and etiology were not. In comparison with the very-high-dose group, the risk of death was 3.871 times (95% CI, 1.043 to 14.370 times) higher in the high-dose group (p=0.043) and 9.775 times (95% CI, 2.493 to 38.320 times) higher in the low-dose group (p=0.001), assuming, in both cases, that age, karyotype, French-American-British classification and etiology of acute myeloid leukemia were constant.

Conclusions Consolidation therapy with high-dose cytarabine appears to improve survival in patients with acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of acute myeloid leukemia
* age 18 years or above
* must have been treated with potentially curative therapy

Exclusion Criteria:

* children or age less than 18 years
* palliative therapy

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute myeloid leukemia in adults treated in the University of Sao Paulo between 1978 and 2007
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pedro ED Llacer, MD, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil